CLINICAL TRIAL: NCT06585592
Title: Establishment of Multimodal-multiparametric Progressive Prediction Models for Thyroid Associated Ophthalmopathy
Status: Completed | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Deputy Director, Shanghai Changzheng Hospital
Other Study IDs: TAO3M-1
Record Dates: First submitted 2024-08-29; First posted 2024-09-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Thyroid-Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TAO

SUMMARY:
Thyroid-associated ophthalmopathy (TAO) is an organ-specific autoimmune disease closely related to thyroid disease, which leads the incidence of orbital disease in adults and is the most common cause of diffuse toxic goiter (Graves disease, GD). The clinical manifestations of TAO are complex and varied. In severe cases, it may seriously impair visual function, affect daily life, and even cause corneal ulceration, perforation, and blindness. Therefore, a reasonable and effective treatment plan should be chosen according to the degree of TAO.

The aim of this clinical study is to:

1. Found characteristic changes from baseline to the end of treatment.
2. Identify characteristic changes associated with treatment response.
3. Construct a multimodal and multiparameter prediction model by characteristic changes.

ELIGIBILITY:
Inclusion Criteria:

* According to the Bartley criteria，diagnosed TAO from 2017/1/1 to 2024/3/31
* Moderate to severe patients defined by EUGOGO
* CAS ≥4 (on the 7-item scale) for the study eye
* Completed orbital MRI at our hospital
* Received complete medical treatment and completed assessment at our hospital

Exclusion Criteria:

* Anticipated need for intervention due to sight-threatening complications or other significant and acute deterioration in vision
* History of systemic (eg, oral or IV) steroid use with a cumulative dose equivalent to < 1 g of methylprednisolone for the treatment of TAO.
* Any major illness/condition or evidence of an unstable clinical condition that, in the investigators judgment, will substantially increase the risk to the participant, or confound the interpretation of safety assessments, if they were to participate in the study
* Any other condition that, in the opinion of the investigator, would impair the ability of the participant to comply with the study procedures or impair the ability to interpret data from the participants participation in the study
* Pregnant or lactating
* Any other condition that,would impair the ability of the participant to undergo orbital MRI

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate to severe active TAO patients who received complete medical treatment and completed assessment .
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with overall response | 1 week after the end of treatment
  Overall response
Percentage of participants with overall response | 24 weeks after the end of treatment
  Overall response
Percentage of participants with overall response | 52 weeks after the end of treatment
  Overall response
Percentage of participants with overall response | 104 weeks after the end of treatment
  Overall response

SECONDARY OUTCOMES:
Incidence and characterization of nonserious treatment emergent adverse events (TEAEs) during the treament | during the treament
Change of Serum TRAb from baseline | 52 weeks after the end of treatment
  including TRAb (IU/l)
Change of Serum T3,T4 level from baseline | 52 weeks after the end of treatment
  inculde T3 (nmol/L), T4 (nmol/L)
Change of Serum lipid parameter | 52 weeks after the end of treatment
  including TG (mmol/L), TC (mmol/L), HDL (mmol/L), LDL (mmol/L)
Change of Serum TSH level from baseline | 52 weeks after the end of treatment
  including TSH (mIU/L)
Change of Serum FT3, FT4 level from baseline | 104 weeks after the end of treatment
  including FT3 (pmol/L), FT4(pmol/L)

OTHER OUTCOMES:
Change of extraocular muscle volume and orbital fat volume by MR | 52 weeks after the end of treatment
change of extraocular muscle volume and orbital fat volume by MRI | 4 weeks after the end of treatment
change of extraocular muscle volume and orbital fat volume by MRI | 24 weeks after the end of treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhai L, Luo B, Wu H, Wang Q, Yuan G, Liu P, Ma Y, Zhao Y, Zhang J. Prediction of treatment response to intravenous glucocorticoid in patients with thyroid-associated ophthalmopathy using T2 mapping and T2 IDEAL. Eur J Radiol. 2021 Sep;142:109839. doi: 10.1016/j.ejrad.2021.109839. Epub 2021 Jul 3. PMID 34252869
- [Background] Li Z, Luo Y, Feng X, Zhang Q, Zhong Q, Weng C, Chen Z, Shen J. Application of Multiparameter Quantitative Magnetic Resonance Imaging in the Evaluation of Graves' Ophthalmopathy. J Magn Reson Imaging. 2023 Oct;58(4):1279-1289. doi: 10.1002/jmri.28642. Epub 2023 Feb 13. PMID 36780178
- [Background] Hu H, Chen L, Zhang JL, Chen W, Chen HH, Liu H, Shi HB, Wu FY, Xu XQ. T2 -Weighted MR Imaging-Derived Radiomics for Pretreatment Determination of Therapeutic Response to Glucocorticoid in Patients With Thyroid-Associated Ophthalmopathy: Comparison With Semiquantitative Evaluation. J Magn Reson Imaging. 2022 Sep;56(3):862-872. doi: 10.1002/jmri.28088. Epub 2022 Jan 29. PMID 35092642